CLINICAL TRIAL: NCT07183787
Title: Comparison of Letrozole Versus Danazole for Pain Management of Female Presenting With Endometriosis
Brief Title: Letrozole vs Danazol for Endometriosis-Related Pain: Randomized Trial
Acronym: LET-DAN RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidra Salman (Other)
Responsible Party: Sponsor-Investigator, Sidra Salman, FCPS TRANIEE, Sharif Medical And Dental College, Lahore
Organization: Sharif Medical And Dental College, Lahore (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SMDC/SMRC/79-18
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2019-12

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Letrozole; Danazol

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group trial with two treatment arms. Participants will be allocated to receive either Letrozole or Danazol for management of endometriosis-related pain. Each participant will remain in their assigned arm throughout the study period.
Masking Description: This is an open-label study due to differences in drug formulations. Participants and investigators will know the assigned intervention; outcomes will be measured using validated patient-reported scales to reduce bias."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Letrozole (Experimental): Participants in this arm will receive Letrozole 2.5 mg orally once daily for 12 weeks for management of endometriosis-related pelvic pain.
  Interventions: Drug: Letrozole
- Arm 2: Danazol (Active Comparator): Participants in this arm will receive Danazol 200 mg orally twice daily for 12 weeks for management of endometriosis-related pelvic pain.
  Interventions: Drug: danazol

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5 mg orally once daily for 12 weeks.
  Arms: Arm 1: Letrozole
Drug: danazol — Danazol 200 mg orally twice daily for 12 weeks.
  Arms: Arm 2: Danazol

SUMMARY:
Background:

Endometriosis is a chronic gynecological condition defined by the ectopic presence of endometrial glands and stroma outside the uterine cavity, most commonly diagnosed via laparoscopy. While its exact etiology remains uncertain, a positive family history is considered a significant risk factor. Danazol has historically demonstrated efficacy in alleviating endometriosis-related pain, while letrozole, primarily used in neoadjuvant settings, has recently emerged as a promising alternative. This study aimed to compare the mean reduction in pain scores between letrozole and danazol in women with laparoscopically confirmed endometriosis.

Objective:

To compare the efficacy of letrozole versus danazol in reducing pain scores among women diagnosed with endometriosis.

Material & Methods:

Study Design: Randomized control trial Setting: Department of Obstetrics & Gynaecology, Sharif Medical and Dental Hospital

DETAILED DESCRIPTION:
Introduction:

Endometriosis is defined by the ectopic presence of functional endometrial glands and stroma outside the uterine cavity, most commonly diagnosed via direct laparoscopic visualization (1). Clinical manifestations include dysmenorrhea, dyspareunia, chronic pelvic pain, and infertility-each of which may significantly impair a woman's quality of life (2). It is a chronic, estrogen-dependent inflammatory condition predominantly affecting women of reproductive age, though adolescents may also be affected (3). Its true prevalence remains uncertain due to underdiagnosis and a diagnostic delay averaging nearly a decade, often attributed to normalization of symptoms and missed recognition by primary care providers. Beyond physical symptoms, endometriosis exerts a profound psychosocial and economic burden on affected individuals, their families, and healthcare systems globally (4).

Pathophysiology and Clinical Impact of Ectopic Endometrial Tissue in Endometriosis Ectopic endometrial tissue typically localizes in the dependent regions of the pelvis, such as the posterior and anterior cul-de-sac, uterosacral ligaments, ovaries, and fallopian tubes; however, extra-pelvic involvement is also possible (5). These implants respond to cyclic hormonal stimulation much like eutopic endometrium, undergoing phases of proliferation, secretion, and subsequent shedding. The metabolic by-products especially cytokines and prostaglandins foster a chronic inflammatory milieu characterized by neovascularization, fibrosis, and pain sensitization. Immunologic dysregulation is also implicated, including aberrant T- and B-cell responses, complement system activation, and elevated interleukin-6 (IL-6) levels in affected individuals. These immunoinflammatory mechanisms lead to adhesion formation, anatomic distortion, and chronic pelvic pain which are the hallmark features of the disease (5).

Classification of Endometriosis:

Endometriosis can be classified into three main types based on lesion location. Superficial peritoneal endometriosis is the most common form, characterized by lesions affecting the peritoneum, the thin membrane lining the pelvic cavity. Endometriomas, or ovarian lesions, are dark, fluid-filled cysts ("chocolate cysts") that develop within the ovaries, often resistant to treatment and capable of damaging healthy ovarian tissue. Deeply infiltrating endometriosis extends beneath the peritoneal surface and may involve adjacent pelvic organs such as the bowel or bladder, occurring in approximately 1% to 5% of affected women (6). (Figure 1).

Figure 1: An Illustration that is an overview of the three primary types of endometrioses based on lesion location: superficial peritoneal lesions, ovarian endometriomas, and deeply infiltrating endometriosis.

Comparative Evaluation of Letrozole and Danazol for Pain Reduction in Females with Endometriosis

Despite varied symptoms, endometriosis diagnosis is often delayed due to the absence of reliable non-invasive biomarkers. Current hormone therapies and analgesics offer limited long-term efficacy, as recurrence is common. Letrozole, an aromatase inhibitor, competitively binds to the cytochrome P450 subunit, reducing estrogen biosynthesis and offering a novel approach to managing endometriosis (7). Letrozole, an aromatase inhibitor, has demonstrated effectiveness in reducing endometriosis-related pain without recurrence post-treatment (8). Danazol, a synthetic androgen, suppresses ovarian activity and modulates immune function but has shown inconsistent results in pain management across studies (9). Although hormone therapies such as letrozole and danazol are widely used for symptom management, existing literature reports conflicting evidence regarding their effectiveness in reducing endometriosis-related pain. The present study seeks to answer the research question: "Among females diagnosed with endometriosis, how does the reduction in pain scores with letrozole therapy compare to danazol therapy over a three-month period, and which agent offers more consistent and sustained pain relief to inform standardized treatment protocols?" Addressing this question may improve patient outcomes in management of pain. So, this study aims to compare letrozole with danazol's impact on pain reduction in females with endometriosis, to guide future treatment protocols and update local clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years

Surgically or clinically diagnosed endometriosis

Moderate to severe pelvic pain (NRS ≥ 4 for at least 3 months)

Willing to use effective contraception during the study

Able to provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding

Severe hepatic disease, thromboembolic disorder, or contraindication to study drugs

Use of hormonal therapy within the last 8 weeks

Known hypersensitivity to Letrozole or Danazol

Participation in another clinical trial within the last 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only biologically female participants are eligible, as endometriosis occurs in women.
Enrollment: 60 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in pelvic pain severity (0-10 Numeric Rating Scale) | 12 weeks
  Mean change in pelvic pain scores measured on a 0-10 numeric rating scale; lower scores indicate improvement.

SECONDARY OUTCOMES:
Change in dysmenorrhea severity | 12 weeks
  Change in dysmenorrhea severity recorded on a standardized 0-10 numeric rating scale; lower scores indicate improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Sharif Medical and Dental College, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haqnawaz F, Virk S, Qadir T, Imam S, Rizvi J. Comparison of Letrozole and Clomiphene Citrate Efficacy along with Gonadotrophins in Controlled Ovarian Hyperstimulation for Intrauterine Insemination Cycles. J Reprod Infertil. 2013 Jul;14(3):138-42. PMID 24163798
- [Background] Rasul SG, Yaqub U, Manzoor M, Mubasshar H. Comparison of Letrozole versus Danazol for the pain management of females presented with endometriosis. Annals of King Edward Medical University. 2017;23(4):514-8.
- [Background] Mehmud G, Akhtar T, Sadia S. Endometriosis: frequency and correlation between symptomatology and disease stage. J Coll Physicians Surg Pak. 2007 Apr;17(4):199-202. PMID 17462175
- [Background] García E, Cruz OP. Regulation of Inflammation Pathways and Inflammasome by Sex Steroid. Reproduction and the Inflammatory Response. 2022:607539061.
- [Background] Khashchenko EP, Uvarova EV, Fatkhudinov TK, Chuprynin VD, Asaturova AV, Kulabukhova EA, Vysokikh MY, Allakhverdieva EZ, Alekseeva MN, Adamyan LV, Sukhikh GT. Endometriosis in Adolescents: Diagnostics, Clinical and Laparoscopic Features. J Clin Med. 2023 Feb 20;12(4):1678. doi: 10.3390/jcm12041678. PMID 36836214
- [Background] Arafah M, Rashid S, Akhtar M. Endometriosis: A Comprehensive Review. Adv Anat Pathol. 2021 Jan;28(1):30-43. doi: 10.1097/PAP.0000000000000288. PMID 33044230